CLINICAL TRIAL: NCT00724672
Title: Whole Human Genome Oligo Microarray Analysis of the Peripheral Blood Mononuclear Cells of Patients With Rheumatoid Arthritis During Different Forms of Anti-Tumor Necrosis-Alpha Treatments.
Brief Title: A Study of Immune Cells in Patients With Rheumatoid Arthritis During Different Types of Anti-TNF Alpha Treatments (Study P05521)
Status: Withdrawn | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05521
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Infliximab; Adalimumab

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- ETA: RA patients who were scheduled to receive etanercept 50 mg subcutaneously once weekly
  Interventions: Drug: etanercept
- IFX: RA patients who were scheduled to receive infliximab 3 mg/kg IV at Weeks 0, 2, and 6
  Interventions: Drug: infliximab
- ADA: RA patients who were scheduled to receive adalimumab 40 mg subcutaneously biweekly
  Interventions: Drug: adalimumab
- non-diseased controls: Healthy individuals who contributed their RNA/cDNA samples prior to the study and for whom ethical approval has already been obtained.

INTERVENTIONS:
Drug: etanercept — etanercept 50 mg subcutaneously once weekly
  Other Names: Enbrel®
  Groups: ETA
Drug: infliximab — infliximab 3 mg/kg IV at Weeks 0, 2, and 6
  Other Names: Remicade®, SCH 215596
  Groups: IFX
Drug: adalimumab — adalimumab 40 mg subcutaneously biweekly
  Other Names: Humira®
  Groups: ADA

SUMMARY:
This 14-week study will observe the gene expression of certain immune cells in patients with rheumatoid arthritis who receive etanercept, infliximab, and adalimumab. Patients at the National Institute of Rheumatology and Physiotherapy, Budapest, who are already scheduled to receive an anti-TNF agent will be asked to participate in this study. Patients will receive their treatment (etanercept, infliximab, or adalimumab) as scheduled, and have blood samples collected during the study and analyzed by the laboratory. Patient's response to their treatment will also be studied based on x-rays and other examinations.

DETAILED DESCRIPTION:
Only patients who - regardless of this study - are scheduled and permitted to receive anti-TNF-alpha treatment because of their RA will be asked to participate. No patient will be recruited only for the sake of the study. The prescribing physicians will not be influenced by the study as to what form of anti-TNF-alpha therapy they should select.

ELIGIBILITY:
Inclusion Criteria:

* Must have active RA (DAS28 >5.1)
* Must have x-ray evidence of an erosive disease,
* Must be eligible for but have never received any anti-TNF treatment,
* Must fulfill the 1987 criteria of the American College of Rheumatology classification criteria for a diagnosis of RA, for at least 3 months,
* Must have failed standard therapy (methotrexate or leflunomide).

Exclusion Criteria:

* Must not be a women who is pregnant or breastfeeding,
* Must not have a history of any malignancy,
* Must not have an active infection,
* Must not be prone to infection,
* Must not have tuberculosis, hepatitis B, hepatitis C, or HIV,
* Must not have septic arthritis of a native prosthetic joint within the last 12 months,
* Must not have NYHA grade 3 or 4 heart failure,
* Must not have a history of demyelinating disease or systemic lupus erythematosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from a single center at the National Institute of Rheumatology and Physiotherapy, Budapest, the largest center for biological therapy in Hungary. Subjects will be patients who are scheduled and permitted to receive anti-TNF-alpha treatment due to their rheumatoid arthritis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Gene expression (under- or overexpression) in the peripheral blood mononuclear cells | Weeks 0, 4, and 14.

SECONDARY OUTCOMES:
Disease Activity measured by DAS28 | Weeks 0 and 14